CLINICAL TRIAL: NCT05275465
Title: A Randomized, Placebo-controlled, Single-Ascending Dose Phase Ia Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HH-006 in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HH-006 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HH006-101
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-006 (Experimental)
  Interventions: Drug: HH-006
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HH-006 — Different dose levels of HH-006
  Arms: HH-006
Drug: Placebo — Different dose levels of placebo
  Arms: Placebo

SUMMARY:
Huahui Health is developing a treatment for Hepatitis B virus. This study is designed to evaluate the safety and tolerability of HH-006, a hepatitis virus neutralizing monoclonal antibody in healthy volunteers, and to determine its pharmacokinetic profile and immunogenicity.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, Phase Ia study aimed to evaluate the safety and tolerability of HH-006 after single ascending doses given as subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male or female individuals aged between 18 to 65 years old
* A bodyweight ≥ 45 kg and the body mass index (BMI) is between 18 to 32 kg/m2.

Exclusion Criteria:

* History of anaphylaxis or other significant allergy in the opinion of the Investigator or known allergy or hypersensitivity to any of the components of the IP
* History of drug, alcohol, or substance abuse
* Any history of liver disease or known hepatic, or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Any history of anaphylaxis, severe allergic reaction, neutralizing antibody generations, or hypersensitivity to albumin or any protein-based therapeutics such as natalizumab (Tysabri) or any other monoclonal antibodies
* Any previous exposure to chimeric, humanized, or human monoclonal antibody, whether licensed or not
* Medical history of active infection (acute or chronic)
* Any safety concern or personal condition that is inappropriate for the study participation per the Investigator's judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Day 1- Day 113
  An AE that started on or after the first study treatment or that worsened after the first study treatment will be regarded as TEAEs.
Severity of treatment emergent adverse events as measured by CTCAE v 5.0 | Day 1- Day 113
Duration of treatment emergent adverse events | Day 1- Day 113

SECONDARY OUTCOMES:
Cmax | Day 1-Day 113
  Maximum observed HH-006 concentration
Tmax | Day 1-Day 113
  Time to maximum observed HH-006 concentration
AUC0- last | Day 1-Day 113
  Area under the plasma concentration-time curve from time zero to the last time point with measurable concentration
AUC0-inf | Day 1- Day 113
  AUC from time zero extrapolated to infinity
t1/2 | Day 1- Day 113
  Apparent terminal half-life
CL (SAD) | Day 1-Day 113
  Apparent total body clearance
CL/F (SAD) | Day 1-Day 113
  Apparent clearance
Vz/F (SAD) | Day 1-Day 113
  Apparent terminal volume of distribution
Titres of anti drug antibodies (ADA) to HH-006 | Day 1- Day 113
  To determine the immunogenicity of HH-006

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, Principal Investigator — Nucleus Network
Locations (1):
- Q-Pharm Pty Ltd (Nucleus Network Pty Ltd), Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No